CLINICAL TRIAL: NCT00002999
Title: S9715, Study of Patients With Advanced Nasopharyngeal Cancers Treated With Chemo-Radiotherapy, Phase II
Brief Title: S9715, Chemotherapy and Radiation Therapy in Treating Patients With Advanced Cancer of the Nasopharynx
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Laurence H. Baker, D.O., Southwest Oncology Group-Group Chair's Office
Purpose: Treatment
Other Study IDs: CDR0000065552; U10CA032102 (NIH); S9715 (Other: SWOG)
Record Dates: First submitted 1999-11-01; First posted 2004-07-05 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Cancer
Keywords: stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Nasopharyngeal Neoplasms | interventions — Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug and combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus radiation therapy in treating patients with advanced cancer of the nasopharynx.

DETAILED DESCRIPTION:
OBJECTIVES: I. Gather additional information and experience regarding the preferred treatment from clinical trial SWOG-8892, chemoradiation for patients with advanced nasopharyngeal cancers (NPC). II. Evaluate survival and progression-free survival and patterns of tumor failure in this new group of patients. III. Assess severe or lethal toxicities that may be encountered after this regimen is employed more widely. IV. Collect NPC tumor specimens for ongoing and future clinical correlative research.

OUTLINE: Patients receive cisplatin by intravenous infusion on day 1 over a 15-20 minute period. This is repeated every 21 days for the first three initial treatments. Patients also receive radiation therapy once daily five times a week during this cycle of treatment. Approximately three weeks after completion of the above treatment, patients are given cisplatin by intravenous infusion over 15-20 minutes as above but at a lower dose. On the same day as cisplatin infusion, patients receive fluorouracil by continuous intravenous infusion over 24 hours for 4 days in a row. This is repeated every 28 days for a total of 3 treatments. Patients are followed until death.

PROJECTED ACCRUAL: 100 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven nasopharyngeal carcinoma (excluding adenocarcinoma), stage III or IV with no evidence of distant metastatic disease (M0) No lung, bone, or liver metastases as proven within 42 days of registration by: -CT scan or nucleotide study of the chest or chest x-ray -liver and bone scan if alkaline phosphatase is greater than the institutional upper limit of normal (ULN), or if clinically indicated -liver scan if SGOT is greater than the institutional ULN

PATIENT CHARACTERISTICS: Age: Any age Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 75,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 1.6 mg/dL AND/OR Creatinine clearance at least 50 mL/minute Other: Not pregnant or nursing Women/men of reproductive potential must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No previous chemotherapy to the primary site or nodes Endocrine therapy: Not specified Radiotherapy: No previous radiotherapy (except for nonmelanomatous skin cancer outside of the radiation therapy treatment volume) Surgery: No previous surgery to the primary site or nodes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhyi Al-Sarraf, MD, Study Chair — Providence Hospital; George L. Adams, MD, Study Chair — Masonic Cancer Center, University of Minnesota